CLINICAL TRIAL: NCT00730431
Title: A Phase I, Randomized, Placebo-Controlled, Dose-Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics of IDX184 After Oral Administration in Healthy Subjects
Brief Title: Single-Dose Escalation Study of IDX184 in Healthy Volunteers (MK-2355-002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2355-002; IDX-08C-002
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Hepatitis C
Keywords: Hepatitis C, healthy volunteers
MeSH Terms: conditions — Hepatitis C | interventions — IDX184

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (7):
- IDX184 5 mg (Experimental): Healthy participants will be administered a single 5 mg dose of IDX184.
  Interventions: Drug: IDX184
- IDX184 10 mg (Experimental): Healthy participants will be administered a single 10 mg dose of IDX184.
  Interventions: Drug: IDX184
- IDX184 25 mg (Experimental): Healthy participants will be administered a single 25 mg dose of IDX184.
  Interventions: Drug: IDX184
- IDX184 50 mg (Experimental): Healthy participants will be administered a single 50 mg dose of IDX184.
  Interventions: Drug: IDX184
- IDX184 75 mg (Experimental): Healthy participants will be administered a single 75 mg dose of IDX184.
  Interventions: Drug: IDX184
- IDX184 100 mg (Experimental): Healthy participants will be administered a single 100 mg dose of IDX184.
  Interventions: Drug: IDX184
- Placebo (Placebo Comparator): Healthy participants will be administered placebo matching IDX184.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IDX184 — IDX184 supplied as size 3, white opaque capsules containing either 5 mg or 25 mg.
  Arms: IDX184 10 mg; IDX184 100 mg; IDX184 25 mg; IDX184 5 mg; IDX184 50 mg; IDX184 75 mg
Drug: Placebo — Placebo supplied as size 3, white opaque capsules matching IDX184 capsules.
  Arms: Placebo

SUMMARY:
The purpose of this study is to obtain single dose safety and pharmacokinetic (PK) data of IDX184 in humans. No formal hypotheses are to be tested in this study.

ELIGIBILITY:
Inclusion Criteria:

* Participants are in general good health.
* All participants of childbearing potential must have agreed to use a consistent form of an acceptable double-barrier method of birth control

Exclusion Criteria:

* Participant is pregnant or breastfeeding.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2008-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Percentage of participants experiencing serious adverse events (SAEs) | Up to Day 6
Percentage of participants experiencing AEs | Up to Day 6
Percentage of participants experiencing dose-limiting toxicity (DLTs) | Up to Day 6
Percentage of participants experiencing grade 1-4 laboratory abnormalities | Up to Day 6

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Zhou XJ, Pietropaolo K, Chen J, Khan S, Sullivan-Bolyai J, Mayers D. Safety and pharmacokinetics of IDX184, a liver-targeted nucleotide polymerase inhibitor of hepatitis C virus, in healthy subjects. Antimicrob Agents Chemother. 2011 Jan;55(1):76-81. doi: 10.1128/AAC.01101-10. Epub 2010 Nov 8. PMID 21060109